CLINICAL TRIAL: NCT04154111
Title: Theta Burst Stimulation as a Tool to Decrease Drinking in Treatment-seeking Alcohol Users
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00061760; R01AA027705 (NIH)
Record Dates: First submitted 2019-11-04; First posted 2019-11-06 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Alcohol Use Disorder; Alcohol Abuse; Alcohol Dependence; Craving
Keywords: Transcranial Magnetic Stimulation; Brain Stimulation; Treatment; Neuroimaging
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (4):
- Real TBS to the mPFC (Experimental): Thirty sessions of real Theta Burst Stimulation (TBS) will be delivered to the left medial prefrontal cortex (mPFC)
  Interventions: Device: Real TBS to the vmPFC
- Sham TBS to the mPFC (Sham Comparator): Thirty sessions of sham Theta Burst Stimulation (TBS) will be delivered to the left medial prefrontal cortex (mPFC)
  Interventions: Device: Sham TBS to the vmPFC
- Real TBS to the dlPFC (Experimental): Thirty sessions of real Theta Burst Stimulation (TBS) will be delivered to the left dorsolateral prefrontal cortex (dlPFC)
  Interventions: Device: Real TBS to the dlPFC
- Sham TBS to the dlPFC (Sham Comparator): Thirty sessions of sham Theta Burst Stimulation (TBS) will be delivered to the left dorsolateral prefrontal cortex (dlPFC)
  Interventions: Device: Sham TBS to the dlPFC

INTERVENTIONS:
Device: Real TBS to the vmPFC — This will be delivered with the Magventure Magpro system; double blinded
  Arms: Real TBS to the mPFC
Device: Sham TBS to the vmPFC — The MagVenture MagPro system has an integrated active sham that passes current through two surface electrodes placed on the skin beneath the coil.
  Arms: Sham TBS to the mPFC
Device: Real TBS to the dlPFC — This will be delivered with the Magventure Magpro system (double blinded).
  Arms: Real TBS to the dlPFC
Device: Sham TBS to the dlPFC — The MagVenture MagPro system has an integrated active sham that passes current through two surface electrodes placed on the skin beneath the coil.
  Arms: Sham TBS to the dlPFC

SUMMARY:
There is growing interest in the utilization of transcranial magnetic stimulation (TMS) as a novel, non-pharmacologic approach to decreasing alcohol use among treatment-seeking individuals with Alcohol Use Disorder (AUD). The results of this study will be used to determine which of the 2 proposed TMS strategies has a larger effect on drinking behavior (% days abstinent, % heavy drinking days) as well as alcohol cue-reactivity in a 4 month period. These data will pave the way for TMS to be used as an innovative, new treatment option for individuals with AUD.

DETAILED DESCRIPTION:
Alcohol Use Disorder (AUD) is prevalent, devastating, and difficult to treat. The majority of therapeutic approaches to date have relied on pharmaceutical modulation or and/or psychotherapy. With a growing knowledge of the neural circuits that contribute to relapse in AUD, there is an emerging interest in developing a novel, neural-circuit specific therapeutic tool to enhance AUD treatment outcomes. The long term goal of this multidisciplinary research team is to develop an evidence-based brain stimulation treatment protocol which will improve AUD treatment outcomes. The competing neurobehavioral decision systems (CNDS) theory posits that in addiction, choice results from a regulatory imbalance between two decision-making systems (impulsive and executive). These behavioral systems are functionally linked to two discrete frontal-striatal circuits which regulate limbic and executive control. Modulating these competing neural circuits (e.g. either dampening the limbic/impulsive system or amplifying the executive control system) may render alcohol users less vulnerable to relapse. These two frontal-striatal neural circuits - the limbic loop (ventromedial prefrontal cortex (VMPFC)-ventral striatum), and executive control loop (dorsolateral PFC (DLPFC)-dorsal striatum) can be differentially stimulated by theta burst stimulation (TBS), a patterned form of transcranial magnetic stimulation.

Over the past 7 years, through the scaffolding of a National Institute on Alcohol Abuse and Alcoholism (NIAAA) P50 Center and a strong Brain Stimulation Research program, this multidisciplinary group of clinicians and neuroscientists has demonstrated) it is possible to differentially activate these circuits through TMS/Blood-oxygen-level-dependent (BOLD) imaging TBS to the VMPFC decreases orbitofrontal cortex and ventral striatal/accumbens BOLD signal in heavy alcohol users TBS also decreases alcohol cue reactivity in this population and in AUD patients currently enrolled in intensive outpatient treatment, 10 days of TBS to the VMPFC is feasible, well-tolerated, increases 1 and 2 month retention rates, and attenuates limbic brain reactivity to alcohol cues after 1 month. While these studies provide a strong foundation for pursuing a larger multisite trial of TBS, the CNDS theory and other alcohol TMS studies suggests that the DLPLC may also be a fruitful treatment target. In a sham-controlled pilot study the study team recently compared the efficacy of VMPFC TBS to DLPFC TBS, and, to the study team's surprise demonstrated that a single session of DLPFC TBS had a greater effect on the brain response to alcohol cues than VMPFC TBS. To resolve this gap in understanding, the investigator proposes a randomized, double-blind, sham-controlled clinical trial to evaluate the relative efficacy of these 2 strategies as novel tools to improve AUD treatment outcomes (e.g. percent days abstinent up to 4 months after TMS treatment initiation). These outcomes will be measured with urine ethyl glucuronide (ETG) and blood carbohydrate deficient transferrin (CDT) measurements. The study team will also evaluate the effect of these TBS treatments brain reactivity to alcohol cues. The investigator's long-term vision is that TBS would be used as an adjuvant to behavioral treatment, enabling individuals to maximize the likelihood of behavioral change.

180 treatment-seeking men and women recruited from the community at large, will be randomized to receive 15 visits of TMS (2x/day; 3x/week, 20-30 min intersession interval) of either real or sham TBS to the VMPFC or left DLPFC while they are enrolled in the proposed study. Randomization will occur after the participant has been consented and screened for eligibility and prior to the first treatment visit. Real/Sham TBS will be delivered three times per week for a total of 15 TMS visits. Quantitative ETG will be collected daily. Quantitative CDT will be collected monthly throughout the course of the study. Additional assessments and/or brain reactivity to alcohol cues will be measured at the following timepoints: baseline screening visit, MRI visit #1 (before TMS treatment visit 1), TMS treatment visits 1, 6, 11, and 15, MRI visit #2, and at the 3 monthly Follow Up visits. A saliva sample taken for genetic analysis of a specific Brain-derived neurotrophic factor (BDNF) variant will be obtained on enrollment and used to also analyze across these measures and individual outcomes in response to TMS. Building on recent pilot data, the study team will test the hypotheses that for both Strategy 1 & 2, real TBS will improve AUD treatment outcomes significantly more than sham. Analysis will be performed using repeated measures analysis of variance (ANOVA) on change scores from baseline for each visit. The main independent variable in the ANOVA will be time (TMS visits 1, 6, 11, and 15), group (VMPFC vs. DLPFC TBS vs. sham) and their interaction.

Aim 1 (Strategy 1): Modulating the limbic system: VMPFC TBS. The study team will evaluate the effect of VMPFC TBS, relative to sham, on number of days abstinent (primary outcome) and heavy drinking days in 30 day intervals for 4 months. Participants will receive stimulation over the left frontal pole electroencephalogram (EEG)10-20 system: Frontal Pole 1 (FP1). This location has been used in previous studies in alcohol users which demonstrate VMPFC target engagement.

Aim 2 (Strategy 2): Modulating the executive system: DLPFC TBS. The study team will evaluate the effect of DLPFC TBS, relative to sham, on the parameters listed. TBS will be delivered over the left DLPFC EEG 10-20 system: Frontal 3 (F3) as this location has also been validated to reliable result in target engagement by this group.

Exploratory Aim- Baseline alcohol cue reactivity as a mediator of TBS clinical response. The study team will test the hypotheses that individuals with a higher ratio of (DLPFC-striatal)/(VMPFC-striatal) response to alcohol cues will be more likely to have a change in drinking after Strategy 2.

ELIGIBILITY:
Inclusion Criteria

1. Age 21- 75.
2. Meets the DSM V criteria for having a current AUD, determined by DSM-V criteria, using the Structured Clinical Interview for DSM-V.
3. Has an AUDIT score above 8 (such that they are at least Medium Risk drinkers according to criteria).

Exclusion Criteria:

1. Any psychoactive substance use (except marijuana and nicotine) within the last 30 days by self-report.
2. Meets DSM V criteria for schizoaffective disorder. [Note: The inclusion of subjects with affective and anxiety disorders is essential because of the marked frequency of the co-existence of mood and other anxiety disorders among patients with AUD at large.
3. Has current suicidal ideation or homicidal ideation.
4. Is currently taking or initiates a medication known to affect alcohol intake and/or craving (e.g., disulfiram. naltrexone, acamprosate, topiramate). [Note: This exclusionary criterion is for scientific rather than safety or patient comfort reasons].
5. Expects a change in their medical history in the next 6 months that would impair their participation in this study [e.g. expected medical procedure, planned pregnancy, initiation of new medication].
6. Females of childbearing potential who are pregnant (by urine HCG), planning to become pregnant, nursing, or who are not using a reliable form of birth control.
7. Suffers from chronic migraines (more than 50% of the days in a month).
8. Does not meet safety criteria for MRI and TMS
9. Is at elevated risk of seizure (i.e., has a history of seizures, is currently prescribed medications known to lower seizure threshold and has had a change in their medication).
10. Is currently enrolled in another form of treatment for alcohol use disorder (This is for scientific reasons to clarify the role of TMS as a treatment agent)
11. History of traumatic brain injury resulting in hospitalization, loss of consciousness for more than 10 minutes, and/or having ever been informed he/she has an epidural, subdural, or subarachnoid hemorrhage.
12. Not able to read and understand questionnaires, assessments, and the informed consent.
13. Clinical Intake Withdrawal Assessment (CIWA) >5 (to prevent delivering TMS to individuals in withdrawal.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2020-05-26 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Percent days abstinent | Through study completion, up to 4 month follow-up
  These outcomes will be measured with urine ETG and CDT drug screens collected monthly up to 4 months.
Percentage of heavy drinking days | Through study completion, up to 4 month follow-up
  The percentage of heavy drinking days will be measured by timeline follow-back. Individuals will be asked to track their daily alcohol consumption over the course of the study.

SECONDARY OUTCOMES:
Changes in Craving | Baseline visit, 1-4 month follow-ups
  Additional craving assessments will be measured through the study as well to detect any changes in craving for alcohol. The alcohol urge questionnaire will be asked prior to TMS administration and at the follow-up visits. This is a scale based on the individuals craving at that moment on a scale of 1-7.
Neuroimaging outcomes: change in drug cue reactivity as specified by changes in BOLD signal | Baseline visit and 1 month follow-up
  The effect of real vs. sham TBS to the left dlPFC vs. real vs. sham TBS to the left vmPFC as a tool to modulate the brain response to alcohol cues will be measured using functional MRI BOLD signal and comparing the relative brain reactivity to the alcohol cues in the executive circuit and limbic circuit before and after TMS.

CONTACTS AND LOCATIONS:
Overall Officials: Merideth A Addicott, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest School of Medicine, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified participant data will be shared with the NIAAA data Archive. Data to be shared will be treatment arm, demographics, substance use assessment results, and imaging data.
Time Frame: Data will be shared following the processing and analyses of imaging data, up to 6 months after publication.
Access Criteria: Access to the deidentified data will only be through the NIAAA Data Repository, who define the criteria for access.

REFERENCES:
- [Derived] Kinney KR, Kirse HA, Stewart NE, Ip EH, Saldana S, DeMaioNewton HE, Kimber M, Smith HR, Douglas HE, Kiraly DD, Hanlon CA, Addicott MA. Theta Burst Stimulation as a tool to decrease drinking in treatment-seeking alcohol users: study protocol for a randomized, double-blind, sham-controlled clinical trial. Trials. 2025 Nov 10;26(1):487. doi: 10.1186/s13063-025-09093-1. PMID 41214823